CLINICAL TRIAL: NCT04333485
Title: Tuberculosis (TB) Aftermath: a Hybrid Type I Effectiveness-implementation Non-inferiority Randomized Trial in India Comparing Two Active Case Finding (ACF) Strategies Among Individuals Treated for TB and Their Household Contacts
Brief Title: Tuberculosis (TB) Aftermath
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Dr. D.Y. Patil Medical College, Hospital and Research Centre (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: IRB00247239; 1R01AI143748-01A1 (NIH)
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Tuberculosis (TB)
Keywords: Household Contacts; Tuberculosis (TB); Recurrence; Active case finding; India; Hybrid effectiveness-implementation trial
MeSH Terms: conditions — Tuberculosis; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based Active Case Finding (HACF) (Active Comparator)
  Interventions: Other: Home-based Active Case Finding (HACF)
- Telephonic Active Case Finding (TACF) (Active Comparator)
  Interventions: Other: Telephonic Active Case Finding (TACF)

INTERVENTIONS:
Other: Home-based Active Case Finding (HACF) — Existing healthcare workers at the participating NTEP TB units will visit all patient homes at 6 and 12 months post-treatment completion. They will administer a standardized TB symptom screen questionnaire to treated TB cases and their household contacts (HHC). All those who screen positive will have a spot sputum taken at the home for microbiological testing at the TB unit.
  Arms: Home-based Active Case Finding (HACF)
Other: Telephonic Active Case Finding (TACF) — Existing healthcare workers at the participating NTEP TB Units will administer a standardized TB symptom screen questionnaire to the index patient via telephone calls at 6 and 12 months post-treatment completion. The index patient will also be asked about any TB symptoms among household contacts (HHCs). If TB is suspected among any HH members, a home visit will be conducted and spot sputum specimens will be collected for microbiological testing at the TB unit.
  Arms: Telephonic Active Case Finding (TACF)

SUMMARY:
TB Aftermath will compare effectiveness, cost-effectiveness and feasibility of two ACF strategies for detecting recurrent TB and provide evidence needed to implement and scale the preferred ACF strategy. The specific aims are:

Primary Aim 1: To conduct a non-inferiority randomized trial to measure the comparative effectiveness of two potentially implementable ACF strategies within India's National TB Elimination Program (NTEP), conducted by existing NTEP healthcare workers (HCWs): (i) home-based ACF (HACF) and (ii) telephonic ACF (TACF).

Primary Aim 2: To characterize implementation processes of the ACF strategies using the Reach, Effectiveness, Adoption, Implementation, and Maintenance (RE-AIM) framework to inform future scale-up and sustainability.

Primary Aim 3: To model the impact and cost effectiveness of the ACF strategies evaluated in the trial, and of potential alternative strategies for the targeting and timing of those strategies.

Secondary Aim: To measure the association of the severity, chronicity and progression of post-TB lung impairment with recurrent TB disease.

DETAILED DESCRIPTION:
Approximately 7% of all reported tuberculosis (TB) cases each year are recurrent, occurring among people who have had TB in the recent or distant past. TB recurrence is particularly common in India, which has the largest TB burden worldwide. Although patients recently treated for TB are at high risk of developing TB again, evidence around effective active case finding (ACF) strategies in this population is scarce. The investigators will conduct a hybrid type I effectiveness-implementation non-inferiority randomized trial to compare the effectiveness, cost-effectiveness, and feasibility of two ACF strategies among individuals who have completed TB treatment and the household contacts (HHCs).

The investigators will enroll 1076 adults (≥ 18 years) who have completed TB treatment at a public TB unit (TU) in Pune, India, along with the HHCs (averaging two per patient, n = 2152). Participants will undergo symptom-based ACF by existing healthcare workers (HCWs) at 6-month intervals and will be randomized to either home-based ACF (HACF) or telephonic ACF (TACF). Symptomatic participants will undergo microbiologic testing through the program. Asymptomatic HHCs will be referred for TB preventive treatment (TPT) per national guidelines. The primary outcome is rate per 100 person-years of people diagnosed with new or recurrent TB by study arm, within 12 months following treatment completion. The secondary outcome is proportion of HHCs < 6 years, by study arm, initiated on TPT after ruling out TB disease. Study staff will collect socio-demographic and clinical data to identify risk factors for TB recurrence and will measure post-TB lung impairment. In both arms, an 18-month "mop-up" visit will be conducted to ascertain outcomes. The investigators will use the RE-AIM framework to characterize implementation processes and explore acceptability through in-depth interviews with index patients, HHCs and HCWs (n = 100). Cost-effectiveness will be assessed by calculating the incremental cost per TB case detected within 12 months and projected for disability-adjusted life years averted based on modeled estimates of morbidity, mortality, and time with infectious TB.

This novel trial will guide India's scale-up of post-treatment ACF and provide an evidence base for designing strategies to detect recurrent and new TB in other high burden settings.

ELIGIBILITY:
Inclusion Criteria:

* Those who are registered at one of the study TB Units (TUs) in Pune district as treatment completed or cured (regardless of type of TB or duration of treatment).
* Confirmed treatment completion or cure status by the referring medical officer of the study TU.
* Date of treatment completion within 60 days of date of enrolment.
* Ability and willingness of participant or legal guardian/representative to provide informed consent to participate in the home-based ACF (HACF) or telephonic ACF arm (TACF).

(NOTE: Illiterate participants or participants with cognitive disabilities may be enrolled based on local regulatory policies, with the appropriate provisions for informed consent.)

- All household contacts of TB cases who are able and willing to provide informed consent to participate are eligible. Household contacts who are <18 years old are eligible for enrolment if a legal guardian/representative provides informed consent.

Exclusion Criteria:

* Completed anti-TB treatment at a private sector clinic or TU outside of the study (final visit not registered at one of the study TB units)
* Actively on anti-TB treatment

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3094 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Rate per 100 person-years of people diagnosed with new or recurrent TB by study arm. | Within 12 months following index TB patient's treatment completion date.
  TB disease will be diagnosed as microbiologically confirmed (positive acid fast bacilli smear or positive Xpert® Mycobacterium tuberculosis/resistance to rifampin (MTB/RIF) assays or positive culture) or clinically diagnosed (initiated on TB treatment with no microbiological confirmation).

SECONDARY OUTCOMES:
Proportion of eligible household contacts (HHCs) <6 years of age, by study arm, initiated on TB preventive treatment (TPT) after ruling out active TB disease. | Up to 18 months following index TB patient's treatment completion date.
  At enrolment, participants will report names of HHCs < 6 years of age and their history of TPT. Children who have not yet initiated TPT will be the denominator and children who initiate TPT following index patient enrolment will be the numerator.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Golub, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Dr. D.Y. Patil Medical College, Hospital and Research Centre, Pune, Maharashtra, India

REFERENCES:
- [Derived] Cox SR, Kadam A, Atre S, Gupte AN, Sohn H, Gupte N, Sawant T, Mhadeshwar V, Thompson R, Kendall E, Hoffmann C, Suryavanshi N, Kerrigan D, Tripathy S, Kakrani A, Barthwal MS, Mave V, Golub JE; TB Aftermath study team. Tuberculosis (TB) Aftermath: study protocol for a hybrid type I effectiveness-implementation non-inferiority randomized trial in India comparing two active case finding (ACF) strategies among individuals treated for TB and their household contacts. Trials. 2022 Aug 5;23(1):635. doi: 10.1186/s13063-022-06503-6. PMID 35932062